CLINICAL TRIAL: NCT00115570
Title: Efficacy and Safety of Insulin Glulisine Compared With Insulin Lispro in Children and Adolescents With Type 1 Diabetes Mellitus: A 26 Week, Multicenter, Open, Parallel Clinical Trial
Brief Title: Comparison of the Ability of Glulisine With Lispro to Control Type 1 Diabetes Mellitus in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6096; HMR 1964
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes,Insulin-Dependent, pediatric,rapid acting injection
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — insulin glulisine; Insulin Lispro; Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Glulisine (Experimental): Insulin Glulisine (100UI/ml), at least twice daily, in association with basal insulin therapy (NPH insulin or insulin glargine for a maximum of 26 weeks
  Interventions: Drug: Insulin glulisine; Drug: insulin glargine; Drug: NPH insulin
- Insulin Lispro (Active Comparator): Insulin Lispro (100UI/ml) Subcutaneous (SC) injection , at least twice daily, in association with basal insulin therapy (NPH insulin or insulin glargine ) for a maximum of 30 weeks
  Interventions: Drug: insulin lispro; Drug: insulin glargine; Drug: NPH insulin

INTERVENTIONS:
Drug: Insulin glulisine — Subcutaneous injection
  Other Names: apidra
  Arms: Insulin Glulisine
Drug: insulin lispro — Subcutaneous injection
  Arms: Insulin Lispro
Drug: insulin glargine — Subcutaneous injection once daily
Drug: NPH insulin — subcutaneous injection twice daily

SUMMARY:
The purpose of this study is to determine if insulin glulisine (Apidra) is as safe and effective a rapid acting insulin as insulin lispro (Humalog) in children and adolescents with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Girls/boys, 4-17 years, inclusive;
* Girls not yet of childbearing potential or, if sexually active, agree to use reliable medically accepted contraceptive measure during study;
* Type 1 diabetes mellitus established in medical history: for example, but not limited to, clear signs of insulinopenia (polyuria, polydipsia, polyphagia, weight loss, ketonuria, ketoacidosis); or glutamic acid decarboxylase (GAD) antibody indicative of type 1 diabetes measured at any time before study; or requiring continuous insulin therapy from time of diagnosis;
* Onset of diabetes at least 1 year prior to visit 1 (V1) of study;
* Uninterrupted insulin therapy for at least 1 year before V1 of study;
* At V1, on stable insulin regimen of either NPH or insulin glargine as basal insulin and willing to have multiple daily injections of insulin;
* Glycated hemoglobin at V1 between ≥ 6.0 and ≤11.0 %;
* Ability/willingness to do blood glucose monitoring using sponsor-provided glucometer and subject diary.

Exclusion Criteria:

* Active proliferative diabetic retinopathy, defined by application of focal or panretinal photocoagulation or vitrectomy, 6 months before V1, or any other unstable/rapidly progressing retinopathy requiring surgical treatment (including laser photocoagulation) during study;
* Diabetes other than type 1 diabetes mellitus;
* Pregnancy (positive pregnancy blood test at V1) or breastfeeding;
* Pancreatectomized subjects;
* Subjects who have had pancreas and/or islet cell transplants;
* Treatment with any anti-diabetic oral agent at any time from diabetes diagnosis;
* Treatment with systemic corticosteroids in last month before V1;
* Subjects on pump therapy during last 2 months before V1;
* Subjects requiring excessively high doses of insulin ("resistant" patients), for example, but not limited to, subjects receiving over 150 IU per day;
* Likelihood of needing treatment during study period with drugs not permitted by protocol
* Treatment with any investigational drug in last month before V1;
* History of primary seizure disorders;
* History of severe hypoglycemic episode accompanied by seizure and/or coma or diabetic ketoacidosis leading to hospitalization, or to care in emergency ward, 3 months prior to V1;
* History of hypoglycemia unawareness;
* History of hypersensitivity to insulin or insulin analogs or any of the excipients in insulin glulisine formulation or any of the excipients in other study insulin preparations formulations;
* Clinically relevant hepatic, neurologic, endocrine, active cancer, or other major systemic disease making implementation of protocol or interpretation of study results difficult and would, in the opinion of the investigator, preclude safe participation of subject in protocol;
* History of cardiac abnormalities and/or cardiovascular disorders;
* History of drug/alcohol abuse;
* Impaired hepatic function shown by, but not limited to, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than twice the normal upper limit for age at V1;
* Impaired renal function shown by, but not limited to, serum creatinine greater than 1.5 times upper limit for age at V1;
* Non fasting triglyceride level of >500 mg/dL (5.7 mmol/L) at V1;
* Parent/legally authorized representative unable to understand nature, scope, possible consequences of study;
* Parent/legally authorized representative unable to read/write;
* Subjects unlikely to comply with protocol, e.g. inability/unwillingness to participate in adequate training, uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing study;
* Children/relatives of employee of sponsor or of sponsor representatives;
* Children or relatives of investigator, any sub-investigator, research assistant, pharmacist, study coordinator or other staff directly involved in conduct of protocol;
* Subjects who have previously been treated with insulin glulisine.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 572 (Actual)
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in total glycated hemoglobin measured as HbA1c equivalents (GHb )from baseline to endpoint | week 26 or last observed treatment

SECONDARY OUTCOMES:
Change from Baseline in GHb at weeks 12 and 26 | weeks 12 and 26
Change from Baseline in Self-monitored glucose parameters | weeks 4, 12, 18, 26, and endpoint;
Incidence of Symptomatic hypoglycemia | first dose of study up to last dose
Change from Baseline in basal insulin dose | week 4, 12, 18, 26, and endpoint;

CONTACTS AND LOCATIONS:
Overall Officials: Dr Arethi PHILOTHEOU, Principal Investigator — UCT Diabetes Clinical Trials Unit - Faculty of Health Sciences - South-Africa
Locations (1):
- Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States